CLINICAL TRIAL: NCT00601133
Title: Quantitative and Clinical Description of Postural Instability in Patient Who Underwent Acute Inpatient Rehabilitation and at Follow-Up
Brief Title: Function and Balance for Inpatient Rehabilitation
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0799
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; Acute Inpatient Rehabilitation; Postural Instability; Balance; Function; Walking; Questionnaire; Survey
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient Postural Instability: Participants having difficulty walking and with balance after cancer treatment that are leaving the M.D. Anderson rehabilitation hospital or after treatment through the rehabilitation mobile team.
  Interventions: Other: Walking Test; Other: Balance Test; Behavioral: Questionnaire; Behavioral: Diary

INTERVENTIONS:
Other: Walking Test — Timed Test 1: From sitting position walk 10 feet quickly, return to sitting position Timed Test 2: Walk 25 feet, turn around, and walk back
  Tests conducted twice, once on departure from rehabilitation center, and again at a return visit 1 month later
Other: Balance Test — Machine balance test: Stand on a platform with a rail, shift weight and try to maintain balance and center of gravity; Results displayed.
Behavioral: Questionnaire — To be completed when leaving the rehabilitation program and again at the study visit 1 month later, lasting about 5 minutes.
  Other Names: Survey
Behavioral: Diary — Record any physical exercise done from departure of rehabilitation center to return visit 1 month later; includes exercises; approximately 5 minutes per entry
  Other Names: journal

SUMMARY:
Objectives:

Primary Objectives:

To determine the change in functional tests of postural control of cancer patients who have completed acute inpatient rehabilitation or complete rehabilitation through mobile team from discharge at 21-60 days (+/- 3) after discharge.

Secondary Objectives:

To assess the correlations between the functional tests of postural control, the balance test and the amount of exercise per week.

DETAILED DESCRIPTION:
To be enrolled in this study, you must be able to walk with or without an assistant device (such as a cane or a walker).

Study Procedures:

If you are found to be eligible to take part in this study, you will do a combination of walking and balance tests twice, once on the day you leave the rehabilitation center or hospital, and again at a return visit 21-60 days (+/-3) later. For the first test, you will get up from a chair and walk 10 feet as quickly, but as safely, as possible. You will then return to the chair and sit again. For the second test, you will walk 25 feet, turn around, and walk back to the starting point as fast and as safely as you can. Both tests will be timed by the study staff.

You will also do a balance test on a machine. You will stand on a platform with a rail to hold on to. You will shift your weight and try to keep your balance and center of gravity, which will be shown on a screen.

You will be given a diary to record any physical exercise you are doing from the time you leave the rehabilitation center to your return visit 21-60 days (+/-3) later. You will be asked to record what kind of exercises (home exercise, home health therapy, or outpatient therapy treatment) you do and for how many hours. It should take about 5 minutes to fill out the diary each time.

You will complete a questionnaire that asks you about your symptoms, such as pain. You will complete it when you leave the rehabilitation program and again at the study visit 21-60 days (+/-3) later. It should take about 5 minutes to complete the questionnaire.

Length of Study:

You will be off study after you complete the second questionnaire.

This is an investigational study.

Up to 58 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, or the legal guardians of patients, must have the ability to understand and willingness to sign a written informed consent document.
2. Patients must be able to ambulate with or without assistant device, without assistance from a person.
3. Patients must have undergone acute inpatient rehabilitation at MDACC or undergone rehabilitation through mobile team.

Exclusion Criteria:

1. Patients who decline to participate or who are determined incapable of completing the research.
2. Active CNS disease, such as clinically-evident metastases or leptomeningeal disease, dementia, or encephalopathy.
3. Patient who is not willing or able to come back for 4+/-1 week routine follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have completed acute inpatient rehabilitation at MDACC
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Patient Results of functional tests of postural control (Timed 50 feet walk + Timed Get Up & Go Test) | Observation points at baseline (discharge) and at post discharge week 4 +/- 1

CONTACTS AND LOCATIONS:
Overall Officials: Ying Guo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org